CLINICAL TRIAL: NCT00343057
Title: Influence of a Simple Information Booklet on the Evolution of Acute Low Back Pain (LBP): a Quasi-experimental Study in a Primary Care Setting.
Brief Title: DISCO - Influence of a Simple Information Booklet on the Evolution of Acute Low Back Pain (LBP)
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Other Study IDs: IXP0001A_9001
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Acute Low Back Pain

INTERVENTIONS:
Other: Patients' questionnaire

SUMMARY:
To assess the impact of standardized written information on outcome in acute LBP.

DETAILED DESCRIPTION:
A 3-month prospective, controlled study with a quasi-experimental design (i.e., a nonrandomized controlled sample with geographic stratification [30 areas]). Control and intervention areas ARE selected for their similarities in rural-to-urban distribution of the population and patients' access to GPs and to minimize risk of overlap between areas.

ELIGIBILITY:
Inclusion Criteria:

* Each GP have to enroll up to 4 patients with acute LBP.

Exclusion Criteria:

Patients are excluded if they

1. are less than 18 years old;
2. have pain for more than 4 weeks;
3. have pain intensity for the previous 24 hours less than 3 on a 11-point numeric scale (0= no pain, 10=maximal pain);
4. have sciatica;
5. have had a previous episode of acute LBP during the last 12 months;
6. have no occupational activities;
7. have consulted another practitioner for the same episode of back pain;
8. are pregnant;
9. have back pain related to infection, tumor, or inflammatory disease; or (j) have previously undergone back surgery.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with acute common low back pain.
Sampling Method: Probability Sample
Enrollment: 2830 (Actual)
Dates: Start 2003-09; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COUDERC, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France

REFERENCES:
- [Derived] Coudeyre E, Tubach F, Rannou F, Baron G, Coriat F, Brin S, Revel M, Poiraudeau S. Effect of a simple information booklet on pain persistence after an acute episode of low back pain: a non-randomized trial in a primary care setting. PLoS One. 2007 Aug 8;2(8):e706. doi: 10.1371/journal.pone.0000706. PMID 17684553